CLINICAL TRIAL: NCT02462850
Title: A Phase 3 Multi-Center Actual-Use Study on the Safety of CL 108 for the Treatment of Moderate to Severe Acute Pain Associated With Osteoarthritis of the Knee or Hip
Brief Title: A Multi-Center Actual-Use Study on the Safety of CL 108 for the Treatment of Moderate to Severe Acute Pain Associated With Osteoarthritis of the Knee or Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Principal Investigator, Joseph Hazelton, Vice President, Regulatory Affairs, Charleston Laboratories, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCT-006
Record Dates: First submitted 2015-05-22; First posted 2015-06-04 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-02

CONDITIONS: Pain; Nausea; Vomiting
Keywords: Pain; Nausea; Vomiting
MeSH Terms: conditions — Pain; Nausea; Vomiting

ARMS (1):
- CL-108 (Experimental): CL-108 Hydrocodone 7.5 mg, acetaminophen 325 mg, Promethazine 12.5 mg
  Interventions: Drug: CL-108

INTERVENTIONS:
Drug: CL-108

SUMMARY:
The purpose of CLCT-006, a multi-center open-label study, is to evaluate the safety of CL-108 (hydrocodone 7.5 mg/APAP 325 mg, promethazine 12.5 mg) for the treatment of moderate to severe acute pain ("flare") associated with osteoarthritis of the knee or hip under actual conditions of use.

DETAILED DESCRIPTION:
The purpose of CLCT-006, a multi-center open-label study, is to evaluate the safety of CL-108 (hydrocodone 7.5 mg/APAP 325 mg, promethazine 12.5 mg) for the treatment of moderate to severe acute pain ("flare") associated with osteoarthritis of the knee or hip under actual conditions of use.

The study will also endeavor to determine

* the physicians' global evaluation of CL-108 as a treatment for moderate to severe acute pain associated with osteoarthritis of the knee or hip
* the patients' global impression of change in pain after treatment of moderate to severe acute pain associated with osteoarthritis of the knee or hip
* any change in the patient's quality of life after treatment of moderate to severe acute pain associated with osteoarthritis of the knee or hip
* the percentage change in pain intensity after treatment of moderate to severe acute pain associated with osteoarthritis of the knee or hip

ELIGIBILITY:
INCLUSION CRITERIA

Informed consent

* Signed consent obtained at screening prior to any procedures being performed.

Gender

* Male or non-pregnant and non-lactating female. A female of child-bearing potential is eligible to participate in this study if she has a negative urine pregnancy test and is post-menopausal or using an acceptable method of birth control (i.e., hormonal, transdermal, or implanted contraceptives, intra-uterine device, diaphragm, condom, abstinence, or surgical sterilization)

Age

* At least 18 years of age

Diagnosis of OA

* Clinical diagnosis of osteoarthritis of the hip and/or knee (signal joints) based on history and physical findings

Confirmation of OA

* Radiographic evidence of OA of the knee or hip (e.g., joint space narrowing, K-L grades 1-4). [Any X-ray finding or report of an X-ray finding at any time that is indicative of OA of the knee or hip confirms the diagnosis of OA.]

Treatment of OA

* Inadequate or unsatisfactory treatment with an NSAID for OA of the knee or hip with no previous use of an opioid for OA (i.e., need for "step up" to opioid treatment).

Flare of OA

* Complaint of acute pain in the knee or hip (i.e., "flare" of osteoarthritis of the knee or hip)

Duration of Acute Pain

* Pain in the signal joint(s) with onset ≤ 14 days

Pain Severity

* Baseline PIS score must be ≥ moderate

Alcohol Intake

* Willing to limit alcohol intake to ≤ 2 drinks per day during the study (i.e., from Screening Visit 1 through Follow-Up Visit 3)

Diary Completion

* Be willing and able to record effectiveness, tolerability, and drug utilization information in the In-Clinic and Outpatient Diaries.

EXCLUSION CRITERIA

Medical Condition

* Presence of a serious uncontrolled medical condition (e.g., poorly controlled hypertension or diabetes)

Confounding Diseases

* Presence of other major joint or bone disease (e.g., gout, inflammatory arthritis, Paget's disease), chronic pain syndrome, or fibromyalgia

Surgery

* Patients who have had surgery on the affected joint within the past 6 months, subjects with a prosthesis at the index joint, patients possibly requiring knee or hip arthroplasty or other surgical procedure on the index joint within 3 months following screening

Drug Allergy

* History of hypersensitivity to an opioid drug, promethazine, acetaminophen, or NSAID (such as ibuprofen) or history of a dystonic/dyskinetic reaction to prior antiemetic or anti-psychotic medication

Confounding and Contraindicated Drugs

* Use within 24 hours of Visit 2 of any analgesic (in particular, opioid), anti-emetic, glucosamine, chondroitin sulfate, or any drug contraindicated with hydrocodone, acetaminophen, or promethazine. Use within 4 months of Visit 2 of any intra-articular or oral corticosteroid or hyaluronic acid.

Investigational Drug Use

* Use of any investigational drug within the past 30 days

Participated in Study

* Previous participation in this study

Pregnancy, Lactation

* Women who are pregnant or breast-feeding

Participant Relationship

* Employee of the Principal Investigator, Sub-investigators or Charleston Laboratories or relative of an employee who is directly involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The safety of CL-108 will be evaluated and assessed by questionnaire, when used, for the treatment of moderate to severe acute pain associated with osteoarthritis of the knee or hip. | 24 hours

SECONDARY OUTCOMES:
An assessment of the study medication will be provided as a treatment for osteoarthritis on the Physician's Global Evaluation (PGE) utilizing a poor to excellent scale | 24 hours
The change in arthritic pain since taking study medication over a specific period will be assessed on the Patient Global Impression of Change scale (PGIC) | 24 hours
Patients will complete a standard QOL questionnaire, comprising five dimensions of health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/ depression). | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Charleston Website — http://www.charlestonlabs.com